CLINICAL TRIAL: NCT00562562
Title: A Pilot MRI Study of Osteopathic Manipulative Treatment of Acute Low Back Pain
Acronym: MRI-OMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Osteopathic Heritage Foundations (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15148; 15148
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MOT (Other): Treatment will focus on the thoracolumbar junction, L5, the sacrum, and the pubes. Treatment will primarily utilize two techniques, muscle energy and ligamentous-articular release, but will be tailored to the findings of the individual patient.
  Interventions: Other: osteopathic manipulative treatment

INTERVENTIONS:
Other: osteopathic manipulative treatment — Treatment will focus on the thoracolumbar junction, L5, the sacrum, and the pubes. Treatment will primarily utilize two techniques, muscle energy and ligamentous-articular release, but will be tailored to the findings of the individual patient.

SUMMARY:
This is a pilot project intended to determine the feasibility of detecting soft tissue changes in response to osteopathic manipulative treatment (OMT). MRIs of the lumbar and pelvic regions of low back pain (LBP) patients will be taken once before and at two different time points after OMT. Images obtained will be quantitatively analyzed for changes in the volumes of back muscles and for changes (T2 signals) indicative of activity levels or pathological conditions. Electromyography (EMG) will be used as an independent measure of back muscle activity for comparison with MRI results.

ELIGIBILITY:
Inclusion criteria:

* Adult patients (18-55)
* Patients with LBP with acute symptoms (within last 3 weeks)
* Test positive for lumbar somatic dysfunction

Exclusion criteria:

* History of any spinal injuries/surgeries
* Positive findings of frank neurological signs during physical exam
* Any other orthopedic or neurological impairment
* Unsuitable for MRI imaging:

  * Cardiac pacemaker or defibrillator
  * Severe Claustrophobia
  * Injured by a metallic object that was not removed
  * Cochlear (ear) implants
  * Surgery involving a metallic implant (e.g. knee replacement)
  * Weight more than 300 lbs/136 kg (weight limit for scanner bed)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
MRI T2 signal changes | within 72 hours

SECONDARY OUTCOMES:
MRI anatomic changes and EMG changes | within 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: John N Howell, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States